CLINICAL TRIAL: NCT02323997
Title: Human Papillomavirus-Associated Cervical Neoplasia in Switzerland at the Start of a National Vaccination Programme: Crosssectional Study
Brief Title: Human Papillomavirus in Cervical Cancer and Pre-cancer in Switzerland: The CIN3+Plus Study
Acronym: CIN3+plus
Status: Completed | Type: Observational
Sponsor: University of Bern (Other)
Collaborators: Federal Office of Public Health, Switzerland (Other Government)
Responsible Party: Sponsor
Other Study IDs: CIN3+plus
Record Dates: First submitted 2014-12-18; First posted 2014-12-24 (Estimated); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Cervical Cancer
Keywords: HPV; cervical cancer; human papillomavirus; cervical pre-cancer; cervical neoplasia
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Histologically confirmed CIN3+ lesions, i.e. CIN3, adenocarcinoma in situ and invasive carcinoma of the cervix.
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will investigate the types of HPV in samples from women with cervical pre-cancer and cancer and gather information to help investigate the impact of HPV vaccination in Switzerland.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Participant is literate in German, French, Italian or English.
* Female, aged 18 years or above.
* Histologically confirmed CIN3+ lesions, i.e. CIN3, adenocarcinoma in situ and invasive carcinoma of the cervix.
* Participant resides in the canton Zurich, Geneva, Basel, Baselland, Luzern or Ticino.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with histologically confirmed CIN3+ lesions
Sampling Method: Non-Probability Sample
Enrollment: 767 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Human papillomavirus presence and type | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Low, Principal Investigator — University of Bern, Institute of Social and Preventive Medicine
Locations (10):
- Switzerland (10):
  - Viollier AG, Allschwil, Basel-Landschaft
  - Universitätsspital Basel, Basel
  - Viollier Weintraub SA, Geneva
  - HUG - Hôpitaux Universitaires de Genève, Geneva
  - Kantonsspital Baselland, Liestal
  - Istituto cantonale di patologia, Locarno
  - Kantonsspital Luzern, Lucerne
  - Institute of Pathology Enge, Zurich
  - Institut für klinische Pathologie Medica, Zurich
  - Universitätsspital Zürich, Zurich

REFERENCES:
- [Result] Egli-Gany D, Spaar Zographos A, Diebold J, Masserey Spicher V, Frey Tirri B, Heusser R, Dillner J, Petignat P, Sahli R, Low N; CIN3+plus study group. Human papillomavirus genotype distribution and socio-behavioural characteristics in women with cervical pre-cancer and cancer at the start of a human papillomavirus vaccination programme: the CIN3+ plus study. BMC Cancer. 2019 Jan 30;19(1):111. doi: 10.1186/s12885-018-5248-y. PMID 30700274